CLINICAL TRIAL: NCT04500145
Title: A Randomized Phase III Study of Comparison Between Simultaneous Integrated Boost (SIB) Intensity-modulated Radiation Therapy (IMRT) Versus Routine IMRT/VMAT in LD-SCLC
Brief Title: Simultaneous Integrated Boost vs. Routine IMRT in Limited-stage Small-cell Lung Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zongmei Zhou, Clinical Professor, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CH-L-072
Record Dates: First submitted 2020-08-03; First posted 2020-08-05 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Small-cell Lung Cancer
Keywords: Limited-stage small-cell lung cancer; radiotherapy; simultaneous integrated boost
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SIB-IMRT (Active Comparator): patients received radiotherapy using IMRT or VMAT，60Gy is given to the field of tumor and metastatic lymph nodes and 50Gy given to CR lesion and high-risk area.concurrent or sequential with 4-6 circles of chemotherapy of EP.
  Interventions: Radiation: SIB-IMRT
- routine (Other): patients received IMRT or VMAT，with the prescription of 60Gy/2Gy/30F to the planning tumor volume ，concurrent or sequential with EP chemotherapy
  Interventions: Radiation: routine IMRT

INTERVENTIONS:
Radiation: SIB-IMRT — 60Gy given to the tumor area，50Gy to the CR lesion or high-risk field at the same time
  Arms: SIB-IMRT
Radiation: routine IMRT — patients received IMRT or VMAT，with the prescription of 60Gy/2Gy/30F to the planning tumor volume ，concurrent or sequential with EP chemotherapy
  Arms: routine

SUMMARY:
Thoracic radiotherapy concurrent with chemotherapy stands for the standard regime for limited staged small cell lung cancer. Involved node radiation（INF） replaced elective node irradiation（ENI） as the more popular since several trails compared the two regimes. simultaneous integrated boost IMRT becomes mature with advancing in IMRT and VMAT. The investigator hypothesis that SIB-IMRT can confine the dose for organs at risk to reduce the toxicities compared with routine IMRT in limited disease small-cell lung cancer.

DETAILED DESCRIPTION:
All patients recruited divided into two arms：SIB-IMRT or routine IMRT，in the routine arm，the prescription dose was 60Gy/2Gy/30f，and in the SIB arm ，60Gy was given to the field of the tumor and metastatic lymph nodes，50Gy was given to CR lesion and high-risk prevention. The physical advantages of SIB-IMRT are to reduce the radiation dose of organs that are at risk in the lungs, esophagus, and heart ensuring the adequate dose for tumor area at the same time. The investigators are carrying out this trial to compare the efficacy, safety, side effects, and type of failure of the two radiotherapy techniques, which will provide a new choice and reliable basis for the future dose-segmentation study of limited-stage small-cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years old,KPS≥80
* pathological small cell lung cancer
* staged as limited disease SCLC（contralateral hilar invasion not included）
* receive radiotherapy concurrent or sequential with chemotherapy，if induction chemotherapy，got PR or SD
* no other tumors
* No serious medical diseases and dysfunction of major organs
* understand this study，able to complete the treatment，accept the following up and sign the informed consent
* Contraception in women of childbearing age.

Exclusion Criteria:

* other malignant tumor（historically or simultaneously）curable non-melanoma skin cancer and cervical carcinoma in situ not included
* Uncontrolled heart disease or myocardial infarction within 6 months
* History of mental illness
* Pregnancy or Lactation
* uncontrolled diabetes、hypertension

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2017-07-20 (Actual); Primary Completion 2021-07-20 (Estimated); Study Completion 2021-10-20 (Estimated)

PRIMARY OUTCOMES:
progress-free survival | 2 year
  the rate of patients survival from the treatment to death or progress

SECONDARY OUTCOMES:
overall survival | 2 year
  rate of patients survival in 2 years
local control rate | 2 year
  recurrence rate of local field in 2 years
side-effects | 3-6months after radiation
  the rate of radiation pneumatic、oesophagitis、haematological toxicity

CONTACTS AND LOCATIONS:
Overall Officials: zongmei zhou, PhD, Principal Investigator — national cancer hospital
Locations (1):
- Department of Radiation Oncology, Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China